CLINICAL TRIAL: NCT05186571
Title: Population-based Incidence of Myopericarditis After Messenger Ribonucleic Acid (mRNA) COVID-19 Vaccination in Danish Children 5-11 Years Old
Brief Title: Myopericarditis After Messenger Ribonucleic Acid (mRNA) COVID-19 Vaccination in Children 5-11 Years Old
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Innovation Fund Denmark (Individual); Ministry of Education, Denmark (Other Government)
Responsible Party: Principal Investigator, Ulrikka Nygaard, Primary investigator, Rigshospitalet, Denmark
Other Study IDs: H-20028631_mRNA
Record Dates: First submitted 2022-01-09; First posted 2022-01-11 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Myopericarditis; Myocarditis; Vaccination; Complications; COVID-19 Pandemic; SARS-CoV2 Infection
Keywords: myopericarditis; myocarditis; Vaccination; SARS-CoV2; mRNA vaccination; children
MeSH Terms: conditions — Myocarditis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Pfizer-BioNTech mRNA COVID-19 vaccination — Vaccination in children 5-11 years of age

SUMMARY:
Myopericarditis is a rare complication to messenger ribonucleic acid (mRNA) COVID-19 vaccines, especially in male adolescents and young adults. The risk in children 5-11 years old is unknown. In Denmark, the Pfizer-BioNTech mRNA COVID-19 vaccination was recommended from December 1, 2021 in individuals aged 5-11 years old. We aim to estimate the incidence of myopericarditis in children 5-11 years old after mRNA COVID-19 vaccination among vaccinated individuals based on a nationwide prospective population-based cohort study with detailed clinical phenotyping.

DETAILED DESCRIPTION:
AIM The project seeks to estimate the incidence of myopericarditis in children 5-11 years old after mRNA COVID-19 vaccination.

HYPOTHESIS The incidence of myopericarditis after mRNA COVID-19 vaccination in children 5-11 years old is significantly lower than the incidence in adolescents.

METHOD Prospective nationwide population-based cohort study of all individuals aged 5-11 years hospitalized due to myocarditis and pericarditis after COVID-19 mRNA vaccination in the period December 1, 2021 to February 1, 2022. The setting is a multicenter study including all 18 Danish Pediatric Departments, providing 24 hours emergency service, and in- and out-patient treatment for all Danish inhabitants aged ≤ 17 years. As part of a pediatric nationwide COVID-19 research set-up, all 18 departments have a principal investigator responsible for prospective real-time data collection of vaccine-associated disease.

To calculate the incidence of myopericarditis among Danish individuals 5-11 years old, the number of individuals who have been mRNA COVID-19 vaccinated will be attained from the National COVID-19-vaccine Database at the Statens Serum Institut.

ELIGIBILITY:
Inclusion Criteria: Children 5-11 years old hospitalized due to myocarditis and pericarditis following mRNA vaccination

Exclusion Criteria: Viral or bacterial cause of myopericarditis, or other known cause of myopericarditis

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children 5-11 years old in Denmark who have received mRNA vaccination
Sampling Method: Non-Probability Sample
Enrollment: 350000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Myopericarditis | Within 42 days after the first vaccine dose

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nygaard U, Holm M, Dungu KHS, Matthesen AT, Stensballe LG, Espenhain L, Hartling U. Risk of Myopericarditis After COVID-19 Vaccination in Danish Children Aged 5 to 11 Years. Pediatrics. 2022 Aug 1;150(2):e2022057508. doi: 10.1542/peds.2022-057508. No abstract available. PMID 35585684